CLINICAL TRIAL: NCT01263119
Title: Effect of LY2216684 on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: A Study of LY2216684 and Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12595; H9P-EW-LNCF (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Warfarin; alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Warfarin, LY2216684 + Warfarin (Experimental): Period 1: Single 10-milligram (mg) warfarin oral dose on Day 1; Washout Period of at least 14 days; Period 2: 18-mg LY2216684 oral dose, once daily on Days 1 to 12, with single 10-mg warfarin oral dose coadministered on Day 3.
  Interventions: Drug: Warfarin; Drug: LY2216684

INTERVENTIONS:
Drug: Warfarin — 10-mg warfarin oral dose
Drug: LY2216684 — 18-mg LY2216684 oral dose

SUMMARY:
The purpose of this study is to determine how warfarin might affect LY2216684 and how giving LY2216684 might affect warfarin in the body. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 mass International Units per milliliter [mIU/mL])
* Have body weight >50 kilogram (kg)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling as per the protocol
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* Are cytochrome P450 2C9 (CYP2C9) extensive metabolizers, as determined by genotyping assessment

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2216684, warfarin, or related compounds
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or show evidence of significant active neuropsychiatric disease, or have a history of suicide attempt or ideation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication (including hormonal contraceptives) within 14 days prior to dosing unless deemed acceptable by the investigator and sponsor's medical monitor
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of cytochrome P450 2C19 (CYP2C19) or CYP2C9 within 30 days prior to dosing
* Have donated blood of more than 500 mL within the last month
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to dosing in each period and while resident at the CRU (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any subjects unwilling to adhere to study caffeine restrictions
* Have used any tobacco-containing or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma
* History or presence of significant bleeding disorders; that is, hematemesis, melanena, severe or recurrent epistaxis, hemoptysis, clinically overt hematuria or intracranial hemorrhage
* Subjects with a history of gastrointestinal ulcers or hemorrhage
* Personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations; for example, cerebral hemorrhage, aneurysm, or premature stroke (cerebrovascular accident <65 years of age)
* Self-reported history of increased bleeding from trauma (for example, prolonged bleeding after tooth extraction)
* History of major surgery within 3 months of screening
* Planned surgery within 14 days after the last day of dosing
* International normalized ratio/prothrombin time (INR/PT), or activated partial thromboplastin time (APTT) above the normal reference range at screening
* Positive fecal occult blood examination at screening
* Female subjects with a history of menorrhagia
* Subjects determined to be unsuitable by the investigator for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Warfarin, LY2216684 + Warfarin
Started | 18
Completed | 16
Not Completed | 2
Not completed — Protocol Violation | 2
Period: Period 2
Arm/Group | Warfarin, LY2216684 + Warfarin
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Warfarin, LY2216684 + Warfarin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6
  Multiple | 4
  White | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity (AUC0-∞) of S-Warfarin
Description: Least Squares (LS) geometric mean was based on AUC0-∞ of S-warfarin; calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours post-warfarin administration on Days 1 and 3
Population: The analysis population included participants who received at least 1 dose of warfarin and had evaluable concentration data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 10 mg Warfarin + 18 mg LY2216684 (Test): Period 2: Day -1=participant admission; Days 1 to 12=18-mg LY2216684 oral dose, once daily; Day 3=single 10-mg warfarin oral dose; Day 13=discharge.
- 10 mg Warfarin Alone (Reference): Period 1: Day -1=participant admission; Day 1=single 10-mg warfarin oral dose; Day 11=discharge. Washout Period: at least 14 days between last dose in Period 1 and first dose in Period 2.
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
nanogram*hour per milliliter (ng*hr/mL) | 22200 [19900 to 24700] | 20800 [18700 to 23200]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.07, 90% CI 2-sided [1.00 to 1.13]

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of S-Warfarin
Description: Least Squares (LS) geometric mean was based on Cmax of S-warfarin; calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
nanogram per milliliter (ng/mL) | 633.00 [576.78 to 694.70] | 566.57 [516.06 to 622.02]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.12, 90% CI 2-sided [1.07 to 1.16]

3. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of S-Warfarin
Description: This outcome was measured based on Tmax of S-warfarin on Day 1 of Period 1 when warfarin was administered alone (reference) and on Day 3 of Period 2 when coadministered with LY2216684 (test).
Time Frame: as for outcome 1
Population: The analysis population included participants who had at least 1 dose of warfarin and had evaluable concentration data.
Measure: Median (Full Range); unit: hour (h)
Groups:
- 10 mg Warfarin Alone (Reference): Period 1: Day -1=participant admission; Day 1=single 10-mg warfarin dose; Day 11=discharge. Washout Period: at least 14 days between last dose in Period 1 and first dose in Period 2.
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 15 | 15
hour (h) | 3.00 [1.00 to 5.00] | 3.00 [1.00 to 4.00]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; p = 0.9551, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.50]

4. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity (AUC0-∞) of R-Warfarin
Description: Least Squares (LS) geometric mean was based on AUC0-∞ of R-warfarin; calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: as for outcome 1
Population: The analysis population included participants who had at least 1 dose of warfarin and evaluable concentration data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
ng*h/mL | 43600 [39600 to 48000] | 38000 [34500 to 41800]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.15, 90% CI 2-sided [1.10 to 1.20]

5. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of R-Warfarin
Description: Least Squares (LS) geometric mean was based on Cmax of R-warfarin; calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: as for outcome 1
Population: The analysis population included participants who had at least 1 dose of warfarin and evaluable concentration data.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
ng/mL | 669.25 [607.10 to 737.76] | 592.38 [537.19 to 653.23]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.13, 90% CI 2-sided [1.09 to 1.17]

6. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) of R-Warfarin
Description: This outcome was measured based on Tmax of R-warfarin on Day 1 of Period 1 when warfarin was administered alone (reference) and on Day 3 of Period 2 when coadministered with LY2216684 (test).
Time Frame: as for outcome 1
Population: The analysis population included participants who had at least 1 dose of warfarin and evaluable concentration data.
Measure: Median (Full Range); unit: h
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 15 | 15
h | 3.02 [2.00 to 5.00] | 4.00 [2.00 to 8.00]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Test type: Superiority or Other; p = 0.6094, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.02]

7. Secondary Outcome: Pharmacodynamics: Area Under the Curve of the International Normalized Ratio (AUCINR) of Warfarin
Description: The INR is the ratio of a participant's prothrombin time to a normal (control) sample. AUCINR was calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: Predose, 6, 12, 24, 48, 72, 96, 120, 144 hours post-warfarin administration on Days 1 and 3
Population: The analysis population included participants who had at least 1 dose of warfarin and evaluable concentration data.
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
ratio | 155 [152 to 157] | 149 [147 to 152]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Least Squares (LS) geometric mean was based on pharmacodynamic AUCINR of warfarin; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [1.02 to 1.05]

8. Secondary Outcome: Pharmacodynamics: Maximum Observed International Normalized Ratio (INRmax)
Description: INR is the ratio of a participant's prothrombin time to a normal (control) sample. INRmax was calculated when warfarin was administered alone (reference) on Day 1 of Period 1 and coadministered with LY2216684 (test) on Day 3 of Period 2.
Time Frame: Predose, 6, 12, 24, 48, 72, 96, 120, 144 hours post-warfarin administration on Days 1 and 3
Population: The analysis population included participants who had at least 1 dose of warfarin and evaluable concentration data.
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference)
Number analyzed (Participants) | 16 | 15
ratio | 1.19 [1.15 to 1.24] | 1.14 [1.10 to 1.19]
Statistical Analysis 1: Comparison: 10 mg Warfarin + 18 mg LY2216684 (Test) vs 10 mg Warfarin Alone (Reference); Least Squares (LS) geometric mean was based on pharmacodynamic INRmax of warfarin; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [1.01 to 1.08]

ADVERSE EVENTS:
Groups:
- 18 mg LY2216684 Alone: Period 2: 18-mg LY2216684 oral dose, once daily on Days 1 to 12.
Arm/Group | 10 mg Warfarin + 18 mg LY2216684 (Test) | 10 mg Warfarin Alone (Reference) | 18 mg LY2216684 Alone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 6/18 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg Warfarin + 18 mg LY2216684 (Test) (N=16) | 10 mg Warfarin Alone (Reference) (N=18) | 18 mg LY2216684 Alone (N=16)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days